CLINICAL TRIAL: NCT01222624
Title: Phase I Dose Escalation Study Evaluating the Safety and Tolerability of PankoMab-GEX™ in Patients With Advanced, TA-MUC1 Positive Solid Malignancies Who Are Not Longer Eligible for Standard Therapy
Brief Title: PankoMab-GEX™: Phase 1 Dose Escalation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEXMab25101
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumors
Keywords: advanced solid malignancies
MeSH Terms: interventions — PankoMab-GEX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PankoMab-GEX™, 3-weekly (Experimental): application, q3w
  Interventions: Drug: PankoMab-GEX™
- PankoMab-GEX™, 2-weekly (Experimental): application q2w
  Interventions: Drug: PankoMab-GEX™
- PankoMab-GEX™, weekly (Experimental): application q1w
  Interventions: Drug: PankoMab-GEX™

INTERVENTIONS:
Drug: PankoMab-GEX™
  Other Names: gatipotuzumab

SUMMARY:
Prospective, open label, dose escalating, multicenter, phase I study measuring the safety, tolerability, and pharmacokinetics of PankoMab-GEX™ after intravenous administration in patients with locally advanced or metastatic solid cancers refractory to standard treatment. The effect of PankoMab-GEX™ on the development of antibodies and tumor response was also evaluated.

DETAILED DESCRIPTION:
Male or female patients of age 18 years or older with a histologically-confirmed, tumor-associated mucin 1 (TA-MUC1) positive, measurable or non-measurable solid tumor who had failed standard therapy and for whom no standard therapy was available.

Open-label, non-randomized, inter-patient dose escalation, multi-center study in a 3 + 3 design.

Patients received PankoMab-GEX™ treatment until disease progression or until the treatment was no longer tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and age ≥ 18 yrs
2. Histologically-confirmed TA-MUC1 positive measurable or non-measurable solid tumors according to RECIST criteria who failed standard therapy and for whom no further standard therapy is available (TA-MUC1 positivity assessed by PankoMab-GEX™ staining in immunohistology of the tumor).
3. Failure of standard therapy or non-availability of standard therapy

   * Patients must have received at least 1 standard chemotherapy during the course of the tumor disease
   * All therapies must be completed 6 weeks (therapeutic monoclonal antibodies) or 4 weeks (all other anti-cancer agents) before start of study treatment and patients must have recovered from all prior therapy toxicities to at least CTCAE grade 1
4. Performance status: Eastern Cooperative Oncology Group (ECOG) 0-1 and estimated life expectancy of > 3 months
5. Adequate organ function as assessed by the following laboratory parameters within 14 days prior to study drug application:

   * Bone marrow function: hemoglobin ≥ 100 g/L; white blood cell count (WBC) ≥ 3.0 x 10^9/L; absolute neutrophil count (ANC) ≥ 1.5x 10^9/L; platelet count ≥ 100 x 10^9/L
   * Hepatic: aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 2.5 times upper limit of normal (ULN) (≤ 5 x ULN if hepatic metastases present); bilirubin ≤ 1.5 x ULN; alkaline phosphatase ≤ 5.0 times upper limit of normal (ULN)
   * Renal: Calculated creatinine clearance > 80 ml/min using the Modification of Diet in Renal Disease (MDRD) formula according to Levey 2005: Glomerular filtration rate (GFR) (ml/min/1.73 m²) = 186 x (serum creatinine /0,95)^-1.154 x (age)^-0.203 x (0.742 females) x (1.21 in black patients)
6. Patients of both genders with procreative potential must use effective contraception while enrolled in the study and for at least 6 weeks after the last study drug infusion
7. Written informed consent must be obtained prior to conducting any study-specific procedures

Exclusion Criteria:

1. Antibody-based immunotherapy within 6 weeks and chemotherapy, radiation or other anti-cancer therapies within 4 weeks prior to study enrolment
2. Any investigational agents at the study enrolment
3. Concurrent anti-tumor therapy or concurrent immunotherapy
4. Concurrent systemic steroids except topical (inhaled, topical, nasal), replacement therapy for the last 28 days. Steroids at low and stable dose (up to 20 mg prednisone) given for chronic disease are also permitted
5. History of allergic reactions to previous antibody therapy
6. Major surgery within 4 weeks prior entering the study and/or incomplete recovery from surgery or planned major surgery
7. Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy such as sarcoidosis, lupus erythematosus, rheumatoid arthritis, glomerulonephritis or systemic vasculitis (except autoimmune thyroiditis with only thyroid hormone replacement and stable disease >1 year)
8. Primary or secondary immune deficiency
9. Clinically active infections > CTCAE grade 2
10. Prior allergic reaction to a monoclonal antibody (e.g. Trastuzumab, Cetuximab or Bevacizumab).
11. Active hepatitis B or C; human immunodeficiency virus (HIV) seropositivity
12. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥3 years will be allowed to enter the study.
13. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug including unstable diabetes mellitus, vena-cava-syndrome, chronic symptomatic respiratory disease.
14. Brain metastasis or leptomeningeal involvement
15. Symptomatic congestive heart failure (New York Heart Association [NYHA] 3 or 4); unstable angina pectoris within 6 months prior to enrollment; significant cardiac arrhythmia, history of stroke or transient ischemic attack within 1 year or left ventricular ejection fraction (LVEF) below the institutional range of normal on a baseline multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
16. History of seizures, encephalitis or multiple sclerosis
17. History of deep vein thrombosis and/or thromboembolic events within the past 6 months before entering the study and/or requiring anticoagulation therapy
18. Evidence or history of bleeding diathesis or coagulopathy
19. Active drug abuse or chronic alcoholism
20. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events assessed with the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE], Version 3.0 | Until 28±2 days following the last infusion
  Adverse events coded using Medical Dictionary for Regulatory Activities (MedDRA) version 13.1
Incidence of Treatment-Emergent abnormal clinical laboratory parameters assessed with the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE], Version 3.0 | Until 28±2 days following the last infusion
  Analyzed in local clinical laboratories
Changes in corrected QT interval (QTc) duration | Until 28±2 days following the last infusion
  based on Electrocardiograms (ECG)
Changes of left ventricular ejection fraction (LVEF) | Until 28±2 days following the last infusion
  based on Multiple Gated Acquisition (MUGA) scan or Echocardiogram (ECHO)
Eastern Cooperative Oncology Group (ECOG) Performance Status | Until 28±2 days following the last infusion
  The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale comprises six grades:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Peak Plasma Concentration (Cmax) | Assessment prior to and 2 min before the end of first infusion, 1 hr and 3 hrs after end of first infusion and 24 hrs after start of first infusion, on Day 2, Day 4, Day 7, Day 14, and then prior to and after end of each infusion up to 15 weeks
  PK of PankoMab-GEX™ in patients after single and multiple dose applications
Pharmacokinetics (PK): Minimum Drug Concentration (Cmin) | Assessment prior to and 2 min before the end of first infusion, 1 hr and 3 hrs after end of first infusion and 24 hrs after start of first infusion, on Day 2, Day 4, Day 7, Day 14, and then prior to and after end of each infusion up to 15 weeks
  PK of PankoMab-GEX™ in patients after single and multiple dose applications
Pharmacokinetics (PK):Time to reach Cmax (tmax) | Assessment prior to and 2 min before the end of first infusion, 1 hr and 3 hrs after end of first infusion and 24 hrs after start of first infusion, on Day 2, Day 4, Day 7, Day 14, and then prior to and after end of each infusion up to 15 weeks
  PK of PankoMab-GEX™ in patients after single and multiple dose applications
Pharmacokinetics (PK): Area under the curve (AUC) | Assessment prior to and 2 min before the end of first infusion, 1 hr and 3 hrs after end of first infusion and 24 hrs after start of first infusion, on Day 2, Day 4, Day 7, Day 14, and then prior to and after end of each infusion up to 15 weeks
  PK of PankoMab-GEX™ in patients after single and multiple dose applications
Pharmacokinetics (PK): Apparent terminal serum half-life (t1/2) | Assessment prior to and 2 min before the end of first infusion, 1 hr and 3 hrs after end of first infusion and 24 hrs after start of first infusion, on Day 2, Day 4, Day 7, Day 14, and then prior to and after end of each infusion up to 15 weeks
  PK of PankoMab-GEX™ in patients after single and multiple dose applications
To evaluate any immunogenicity | Anti-drug antibodies (ADAs) were to be measured before the first infusion of study medication, prior to the second infusion, 4 weeks and 8 weeks after the last study medication administration.
  Anti-drug antibodies (ADAs)
Tumor response: Best observed response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Tumors were measured by computed tomography (CT)-scan or magnetic resonance imaging (MRI) and evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Tumor response: Objective response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Tumors were measured by computed tomography (CT)-scan or magnetic resonance imaging (MRI) and evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Tumor response: Clinical benefit rate (CBR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Tumors were measured by computed tomography (CT)-scan or magnetic resonance imaging (MRI) and evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Tumor response: Duration of response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Tumors were measured by computed tomography (CT)-scan or magnetic resonance imaging (MRI) and evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Tumor response: Duration of stable disease | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Tumors were measured by computed tomography (CT)-scan or magnetic resonance imaging (MRI) and evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Glycotope GmbH, Study Director — Glycotope GmbH
Locations (3):
- Glycotope Investigational Site, Hamburg, Germany
- Glycotope Investigational Site, Milan, Italy
- Glycotope Investigational Site, Bellinzona, Switzerland

REFERENCES:
- [Result] Fiedler W, DeDosso S, Cresta S, Weidmann J, Tessari A, Salzberg M, Dietrich B, Baumeister H, Goletz S, Gianni L, Sessa C. A phase I study of PankoMab-GEX, a humanised glyco-optimised monoclonal antibody to a novel tumour-specific MUC1 glycopeptide epitope in patients with advanced carcinomas. Eur J Cancer. 2016 Aug;63:55-63. doi: 10.1016/j.ejca.2016.05.003. Epub 2016 Jun 7. PMID 27285281